CLINICAL TRIAL: NCT06723080
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of VC005 Tablets in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Phase III Clinical Study of VC005 Tablets in Adult Patients With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-302
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Moderate to Severe Atopic Dermatitis
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VC005 low dose group (Experimental)
  Interventions: Drug: VC005 low dose group
- VC005 high dose group (Experimental)
  Interventions: Drug: VC005 high dose group
- VC005 placebo group (Placebo Comparator)
  Interventions: Drug: VC005 Placebo group

INTERVENTIONS:
Drug: VC005 low dose group — VC005 low dose group repeat administration
  Arms: VC005 low dose group
Drug: VC005 high dose group — VC005 high dose group repeat administration
  Arms: VC005 high dose group
Drug: VC005 Placebo group — VC005 Placebo group repeat administration
  Arms: VC005 placebo group

SUMMARY:
This clinical trial is a multicenter, randomized, double-blind, controlled phase III clinical study

ELIGIBILITY:
Inclusion Criteria:

(1）The patient understands and voluntarily signs the Informed Consent Form (ICF), and has the willingness and ability to complete the regular visits,treatment plans, laboratory tests and other experimental procedures required by the program. (2) Male or female patients aged ≥18 and ≤75 years at the time of signing the ICF. (3) Meet Hanifin-Rajka diagnostic criteria at screening and have atopic dermatitis （AD) symptoms for at least 1 year prior to baseline. (4) At screening and baseline, meets criteria for moderately severe AD based on the investigator's assessment of 3 of the following:Eczema area and severity index (EASI) score ≥12;Psoriasis Area Severity Index (IGA) score ≥3;AD involvement in ≥10% of the Body Surface Area (BSA). (5) Recent (within 1 year prior to screening) topical treatment for AD with inadequate or intolerant clinical response, as determined by the investigator

Exclusion Criteria:

(1) Inability to swallow the test drug or refractory nausea and vomiting, malabsorption, extracorporeal biliary shunt, or the presence of a gastrointestinal disorder (e.g., Crohn's disease, ulcerative colitis, or short bowel syndrome) or other malabsorption condition that interferes with the absorption of the drug; (2) Current or history of lymphoproliferative disorders or presence of signs or symptoms suggestive of possible lymphoproliferative disorders of lymphoid tissue, including lymphadenopathy or splenomegaly; malignancies of any kind, or a history of any malignancy within the 5 years prior to Screening (except for completely resected carcinoma in situ of the cervix or non-metastatic squamous cell or basal cell carcinoma of the skin or papillary carcinoma of the thyroid gland); (3) Patients with prior thromboembolism (including deep vein thrombosis, pulmonary embolism, arterial thrombosis, etc.) or other high-risk groups prone to thromboembolism; (4) Patients with a history of herpes virus infection within the last 1 month or those with recurrent episodes of herpes zoster (≥2), disseminated herpes zoster, disseminated herpes simplex, or those for whom herpes zoster or herpes simplex infections cannot be excluded at this time;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving at least a 75% reduction in Eczema Area and Severity Index (EASI 75) from Baseline at Week 16 | week 16

CONTACTS AND LOCATIONS:
Overall Officials: qianjin Lu, Principal Investigator — Chinese Academy of Medical Sciences Hospital of Skin Disease
Locations (1):
- Chinese Academy of Medical Sciences Hospital for Skin Diseases, Nanjing, Jiangsu, China